CLINICAL TRIAL: NCT03948165
Title: Distal Transradial Access for Coronary Angiography and Percutaneous Coronary Intervention: An Observational Study in a Latin-American Centre
Brief Title: Distal Transradial Access for Coronary Angiography and Percutaneous Coronary Intervention.
Status: Completed | Type: Observational
Sponsor: CMN "20 de Noviembre" (Other)
Responsible Party: Principal Investigator, Héctor Hugo Escutia Cuevas, Clinical Professor, CMN "20 de Noviembre"
Other Study IDs: 34.2018
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Coronary Artery Disease
Keywords: dTRA; transradial access; distal; coronary
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Distal Radial Approach: Distal transradial access will be performed on patients above 18 years of age, undergoing diagnostic and/or therapeutic coronary angiography, with palpable pulse at the level of the radial fossa, and these patients will be also subjected to the following tests: Allen maneuver and Barbeau maneuver; a positive Allen test was indication to perform the transradial access, while a type D Barbeau test will be a contraindication for it.
  Interventions: Procedure: Distal Transradial Access

INTERVENTIONS:
Procedure: Distal Transradial Access — The distal radial artery needs to be punctured with specialized equipment with a 20, 21 or 22-gauge puncture needle, using a transfixion or anterior wall technique. A 0.025 in, 46 cm guide was introduced in the system, followed by the introduction of the 5 Fr, 6 Fr, 7Fr hydrophilic arterial sheath or 5 Fr, 6 Fr or 7 Fr Glidesheath Slender introducer (TerumoIS, Tokyo, Japan), after a small incision in the skin.

SUMMARY:
Introduction: The distal radial technique which consists of canalizing the radial artery through the anatomical snuffbox has recently emerged as an alternative arterial intervention for diagnostic and therapeutic coronary catheterization.

Aims: To evaluate the feasibility and safety of the distal transradial approach (dTRA) as a default route for coronary angiography (CAG) and percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
Conventional transradial intervention is now considered the first intention technique for coronary access. The principal advantages are the increase in safety due to the reduction of major bleeding complications, as well as an increase in the patient's comfort due to the immediate post-procedure mobilization.

The safety of conventional transradial catheterization is determined mainly by the favorable anatomical relationship between the radial artery and the adjacent structures. No important vein or nerve is located near the artery, which minimizes the chances of damaging these structures. Due to the superficial trajectory of the radial artery, hemostasis can be easily performed with local compression. Traumatic or thrombotic arterial occlusion does not put the viability of the hand at risk while there is an adequate collateral blood flow from the ulnar artery, or from the interosseous artery.

Among the expected complications and limitations for future interventions is radial artery occlusion, which is estimated to occur in 1-10% of patients undergoing transradial intervention, and it has been considered the "Achilles heel" of transradial intervention for patients who eventually require new coronary interventions due to the complexity of their cardiac disease, because it originates in the sheath insertion site due to endothelial damage, blood flow cessation, and secondary thrombosis, and has an early occurrence after transradial catheterization. The radial artery occlusion is clinically silent due to the blood flow supply through the ulnar artery, which becomes a significant problem just at the time of the study execution, enhancing the interventionist cardiologist to perform a new vascular access.

The distal radial technique, which consists of canalizing the radial artery through the anatomical structure called the snuffbox (anatomical snuffbox, radial fossa, fovea radialis) on the dorsal aspect of the hand, has recently emerged as an alternative arterial intervention for diagnostic and therapeutic coronary catheterization, allowing the conservation of the radial artery for classical transradial intervention in patients who, according to the complexity of their heart disease, require new coronary interventions.

Another important characteristic of this technique is a proximal puncture of the short artery of the thumb and distally to the branch that irrigates the superficial palmar arch. This is because an occlusion at this site maintains anterograde flow towards the superficial palmar arch. This reduces the risk of formation of retrograde thrombus in the proximal radial artery located in the forearm, a frequent finding in patients who develop radial artery occlusion due to traumatic punctures or traumatic hemostasis at the traditional radial puncture site. Flow towards the thumb is maintained by way of the superficial palmar arch, preventing ischemia and disability of the hand.

This technique of distal transradial intervention has been performed in Mexico since 2017. The present research aims to describe the characteristics, complications, and benefits of this procedure carried out on a consecutive series of patients in a Latin-American centre.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old
* Undergoing diagnostic and/or therapeutic coronary angiography
* With palpable pulse at the level of the radial fossa
* With a positive Allen test
* A positive Barbeau test, except type D.

Exclusion Criteria:

* Patients with type D Barbeau test
* cardiogenic shock within the previous 48 hours
* anticoagulation contraindication
* uncontrolled arterial hypertension
* peripheral arterial disease
* proximal radial artery diameter by duplex ultrasound <1.9 mm
* radial access used within the previous 6 weeks
* proximal radial artery occlusion
* refusal of registration admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with radial artery pulse palpable in the radial fossa.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of complications associated with the procedure | 24 hours
  Complications associated with the procedure: haematoma, ecchymosis, bleeding, arterial dissection, thrombosis, radial artery occlusion.

SECONDARY OUTCOMES:
Unsuccessful distal radial artery procedure | 24 hours
  Incidence of arterial crossover

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Muratalla-Gonzalez, MD, Study Chair — CMN "20 de Noviembre"
Locations (1):
- National Medical Centre "November 20", Mexico City, Mexico City, Mexico